CLINICAL TRIAL: NCT04863417
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, VEHICLE-CONTROLLED, PARALLEL COHORT STUDY TO EVALUATE THE SAFETY, TOLERABILITY, SKIN IRRITATION POTENTIAL AND PHARMACOKINETICS OF MULTIPLE-DOSE, TOPICAL ADMINISTRATION OF PF-07038124 TO JAPANESE HEALTHY PARTICIPANTS
Brief Title: Study to Evaluate the Safety, Local and Systemic Tolerability, and Pharmacokinetics of Multiple-Dose Topical Administration of PF-07038124 in Japanese Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3941003
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Results first posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (2000 cm2 Body Surface Area) (Experimental)
  Interventions: Drug: PF-07038124 or vehicle
- Cohort 2 (4000 cm2 Body Surface Area) (Experimental)
  Interventions: Drug: PF-07038124 or vehicle

INTERVENTIONS:
Drug: PF-07038124 or vehicle — PF-07038124 0.01% or vehicle Ointment QD applied to 2000 cm2 Body Surface Area
  Arms: Cohort 1 (2000 cm2 Body Surface Area)
Drug: PF-07038124 or vehicle — PF-07038124 0.01% or vehicle Ointment QD applied to 4000 cm2 Body Surface Area
  Arms: Cohort 2 (4000 cm2 Body Surface Area)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, skin irritation potential, and PK of PF-07038124 in Japanese healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 20 to 55 years of age, inclusive, at the time of signing the ICD.
2. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and 12-lead ECG.
3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
4. Participants must have 4 biologically Japanese grandparents who were born in Japan.
5. BMI of 17.5 to 25 kg/m2; and a total body weight >50 kg (110 lb).
6. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

1. Participants who have any visible skin damage or skin condition (eg, sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations) in or around the application site which, in the opinion of the investigative personnel, will interfere with the evaluation of the test site reaction.
2. Participants who have a history of or have active forms of dermatitides/eczematous conditions (eg, contact dermatitis, seborrhhoeic, discoid, gravitational, asteatotic and dishydrotic eczema) or other inflammatory skin diseases(eg, psoriasis, viral infection, fungal infection, bacterial infection) that would interfere with evaluation of the test site reaction.
3. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
4. History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, HBcAb, HCVAb, or syphilis at screening. Hepatitis B vaccination is allowed.
5. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
6. Acute disease state (unstable medical condition such as nausea, vomiting, fever or diarrhea, etc) within 7 days of Day 1.
7. Have undergone significant trauma or major surgery within 4 weeks of screening.
8. Use of prescription or nonprescription drugs and dietary and herbal supplements within 14 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
9. Previous administration with an investigational drug within 4 months (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
10. A positive urine drug test at screening and/or Day -1.
11. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest.
12. Baseline 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, baseline QTcF interval >450 msec, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second or third degree AV block, or serious bradyarrhythmia's or tachyarrhythmias).
13. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * AST or ALT level ≥1.5 × ULN;
    * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is≤ ULN.
14. A positive COVID-19 test at screening.
15. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
16. Blood donation (excluding plasma donations) of approximately ≥400 mL within 3 months or ≥200 mL within a month prior to dosing. Additionally, approximately ≥400 mL within 4 months for female participants.
17. History of serious adverse reactions or hypersensitivity to any topical drug; or known allergy to any of the study intervention or any components in the study intervention or history of hypersensitivity; or allergic reactions to any of the study preparations.
18. Not willing to refrain from shaving (Note: shaving around face is permitted), the use of depilatories or other hair-removal activities, antiperspirants, lotions, skin creams, fragrances or perfumes, or body oils (eg, baby oil; coconut oil), use of hair products, hair gels, and hair oil in the treatment areas for 48 hours prior to admission to the CRU and for the duration of the stay in the CRU.
19. History of sensitivity to heparin or heparin induced thrombocytopenia only if heparin is planned to flush intravenous catheters.
20. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
21. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- P-one clinic, Keikokai medical corporation, Hachiōji, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Ono R, Wada S, Matsuoka N, Tsunemi Y, Furihata K. Phase 1 Study of Topical Administration of Novel Phosphodiesterase-4 Inhibitor PF-07038124 in Japanese Healthy Participants. J Dermatol. 2025 Nov;52(11):1666-1673. doi: 10.1111/1346-8138.17914. Epub 2025 Aug 17. PMID 40820616
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3941003

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 participants signed the informed consent form (ICF). All were enrolled into the study and randomized to a study treatment. None of them were screen failure.
Groups:
- Cohort 1: PF-07038124 2000 Centimeter Square (cm^2) Body Surface Area (BSA): Participants were randomized to receive PF-07038124 ointment 0.01 percentage (%) for topical application on 2000 cm^2 of skin from Day 1 to Day 10 once daily (QD). The application area was identified by the investigator. Participants were followed up for 28 to 31 days after last dose of study drug.
- Cohort 1: Vehicle 2000 cm^2 BSA: Participants were randomized to receive vehicle ointment for topical application on 2000 cm^2 of skin from Day 1 to Day 10 QD. The application area was identified by the investigator. Participants were followed up for 28 to 31 days after last dose of study drug.
- Cohort 2: PF-07038124 4000 cm^2 BSA: Participants were randomized to receive PF-07038124 ointment 0.01% for topical application on 4000 cm^2 of skin from Day 1 to Day 10 QD. The application area was identified by the investigator. Participants were followed up for 28 to 31 days after last dose of study drug.
- Cohort 2: Vehicle 4000 cm^2 BSA: Participants were randomized to receive vehicle ointment for topical application on 4000 cm^2 of skin from Day 1 to Day 10 QD. The application area was identified by the investigator. Participants were followed up for 28 to 31 days after last dose of study drug.
Period: Overall Study
Arm/Group | Cohort 1: PF-07038124 2000 Centimeter Square (cm^2) Body Surface Area (BSA) | Cohort 1: Vehicle 2000 cm^2 BSA | Cohort 2: PF-07038124 4000 cm^2 BSA | Cohort 2: Vehicle 4000 cm^2 BSA
Started | 4 | 2 | 4 | 2
Completed | 4 | 2 | 4 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of study drug. Participants were analyzed based on the product they received.
Groups:
- Cohort 1: PF-07038124 2000 cm^2 BSA: Participants were randomized to receive PF-07038124 ointment 0.01% for topical application on 2000 cm^2 of skin from Day 1 to Day 10 QD. The application area was identified by the investigator. Participants were followed up for 28 to 31 days after last dose of study drug.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: PF-07038124 2000 cm^2 BSA | Cohort 1: Vehicle 2000 cm^2 BSA | Cohort 2: PF-07038124 4000 cm^2 BSA | Cohort 2: Vehicle 4000 cm^2 BSA | Total
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 12
Age, Customized [Count of Participants; unit: Participants]
  26-35 years | 1 | 1 | 1 | 1 | 4
  36-45 years | 2 | 0 | 1 | 1 | 4
  46-55 years | 1 | 1 | 2 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 4 | 2 | 4 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 4 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 2 | 4 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant temporally associated with the use of study intervention, not necessarily considered related to the study intervention. SAEs were defined as any AE which occurred at any dose and resulted in any of following outcomes: death, life-threatening experience (risk of death at the time of event), required inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly. TEAEs are events between first dose of study drug up to maximum of 31 days after last dose of study drug.
Time Frame: Day 1 up to maximum of 31 days after last dose of study drug (maximum up to 41 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Vehicle: This arm included participants who receive vehicle ointment for topical application on 2000 cm^2 and 4000 cm^2 of skin from Day 1 to Day 10 QD. The application area was identified by the investigator. Participants were followed up to 28 days after last dose of study drug.
Arm/Group | Cohort 1: PF-07038124 2000 cm^2 BSA | Cohort 1: Vehicle 2000 cm^2 BSA | Cohort 2: PF-07038124 4000 cm^2 BSA | Cohort 2: Vehicle 4000 cm^2 BSA | Pooled Vehicle
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4
Participants
  TEAEs | 0 | 0 | 1 | 0 | 0
  SAEs | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs During the Study
Description: Vital signs that were assessed included supine systolic blood pressure, diastolic blood pressure and supine pulse rate. Clinical significance was determined based on investigator's discretion.
Time Frame: Day 1 up to Day 11
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-07038124 2000 cm^2 BSA | Cohort 1: Vehicle 2000 cm^2 BSA | Cohort 2: PF-07038124 4000 cm^2 BSA | Cohort 2: Vehicle 4000 cm^2 BSA | Pooled Vehicle
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4
Participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) During the Study
Description: ECG parameters that were assessed included PR interval, QRS interval, QT interval, QTCF (Fridericia's correction formula) and heart rate. Clinical significance was determined based on investigator's discretion.
Time Frame: Day 1 up to Day 11
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-07038124 2000 cm^2 BSA | Cohort 1: Vehicle 2000 cm^2 BSA | Cohort 2: PF-07038124 4000 cm^2 BSA | Cohort 2: Vehicle 4000 cm^2 BSA | Pooled Vehicle
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Clinical laboratory tests included hematology, clinical chemistry and urinalysis parameters. Clinical significance of abnormalities in these parameters was determined based on investigator's discretion.
Time Frame: Day 1 up to Day 11
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-07038124 2000 cm^2 BSA | Cohort 1: Vehicle 2000 cm^2 BSA | Cohort 2: PF-07038124 4000 cm^2 BSA | Cohort 2: Vehicle 4000 cm^2 BSA | Pooled Vehicle
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4
Participants | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants Categorized According to Draize Scores (Maximum Score) for Local Skin Irritation Assessment During the Study, Regardless of Visit and Assessment Location
Description: Draize score was used to measure the skin irritability based on erythema, edema, papules, and vesicles at the administration site. Draize score ranged from 0 to 4, where 0 indicated no reaction visible, 1 indicated trace reaction (barely perceptible pinkness), 2 indicated mild reaction (readily visible pinkness), 3 indicated moderate reaction (definite redness) and 4 indicated strong to severe reaction (very intense redness). In this outcome measure number of participants are reported according to their maximum score they had during the study through Day 1 to 11, regardless of visit and assessment location.
Time Frame: Through Day 1 to Day 11 (prior to application from Day 1-10 and 24 hours post application on Day 10)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-07038124 2000 cm^2 BSA | Cohort 1: Vehicle 2000 cm^2 BSA | Cohort 2: PF-07038124 4000 cm^2 BSA | Cohort 2: Vehicle 4000 cm^2 BSA | Pooled Vehicle
Number analyzed (Participants) | 4 | 2 | 4 | 2 | 4
Participants
  Score 0 | 4 | 2 | 4 | 2 | 4
  Score 1 | 0 | 0 | 0 | 0 | 0
  Score 2 | 0 | 0 | 0 | 0 | 0
  Score 3 | 0 | 0 | 0 | 0 | 0
  Score 4 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-07038124
Description: AUCtau= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to the time end of dosing interval (24 hours post-dose). AUCtau only for PF-07038124 reporting groups is reported. Participants must have a minimum of 3 quantifiable concentrations to report AUC. All concentrations lesser than lower limit of quantification, then AUCtau=0.
Time Frame: 0 to 24 hours post dose on Day 1 and Day 10
Population: Pharmacokinetic (PK) analysis set included all participants who received at least one dose of PF-07038124 and in whom at least 1 plasma sample concentration value was reported. Here, 'Number Analyzed' signifies participants who had minimum of 3 concentrations to report AUCtau or when all concentrations LLOQ (AUCtau would be 0).
Measure: Geometric Mean (Full Range); unit: Picograms*hour per milliliter
Arm/Group | Cohort 1: PF-07038124 2000 cm^2 BSA | Cohort 2: PF-07038124 4000 cm^2 BSA
Number analyzed (Participants) | 4 | 4
Picograms*hour per milliliter
  Day 1 | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  Day 10: number analyzed (Participants) | 3 | 4
  Day 10 | 0.000 [0.000 to 0.000] | 0.1650 [0.000 to 287]

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-07038124
Description: Cmax only for PF-07038124 reporting groups is reported.
Time Frame: Day 1 and 10: Pre-dose (0 hour), 1, 2, 4, 6, 8 and 12, 24 hours post-dose
Population: PK analysis set included all participants who received at least one dose of PF-07038124 and in whom at least 1 plasma sample concentration value was reported.
Measure: Geometric Mean (Full Range); unit: Picograms per milliliter
Arm/Group | Cohort 1: PF-07038124 2000 cm^2 BSA | Cohort 2: PF-07038124 4000 cm^2 BSA
Number analyzed (Participants) | 4 | 4
Picograms per milliliter
  Day 1 | 0.000 [0.000 to 0.000] | 0.000 [0.000 to 0.000]
  Day 10 | 0.001965 [0.000 to 14.9] | 0.03911 [0.000 to 17.6]

ADVERSE EVENTS:
Time Frame: Day 1 up to maximum of 31 days after last dose of study drug (maximum up to 41 days)
Arm/Group | Cohort 1: PF-07038124 2000 cm^2 BSA | Cohort 1: Vehicle 2000 cm^2 BSA | Cohort 2: PF-07038124 4000 cm^2 BSA | Cohort 2: Vehicle 4000 cm^2 BSA | Pooled Vehicle
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 0/4 | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/4 | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 1/4 | 0/2 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PF-07038124 2000 cm^2 BSA (N=4) | Cohort 1: Vehicle 2000 cm^2 BSA (N=2) | Cohort 2: PF-07038124 4000 cm^2 BSA (N=4) | Cohort 2: Vehicle 4000 cm^2 BSA (N=2) | Pooled Vehicle (N=4)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT04863417/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT04863417/SAP_001.pdf